CLINICAL TRIAL: NCT05828368
Title: Determination of Dickkopf-3 rs11544814 and Complement Factor H rs10737680 Genetic Polymorphism and Change in Their Protein Levels Before and After Non Surgical Periodontal Therapy in Periodontitis Patients With and Without Coronary Artery Disease
Brief Title: DKK-3 rs11544814 and CFH rs10737680 Polymorphism and Protein Levels With Non Surgical Periodontal Therapy in Periodontitis Patients With and Without CAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor department of periodontology, Meenakshi Ammal Dental College and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; Cardiovascular disease; Non surgical periodontal therapy; Biomarker
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Cardiovascular Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP I: 40 systemically healthy subjects with healthy periodontium. (No Intervention): Systemically healthy subjects with healthy periodontium having probing pocket depth (PPD) ≤3mm, no clinical attachment loss (CAL=0) and bleeding on probing ≤ 10% of sites.
- GROUP II: 40 periodontitis patients without coronary artery disease (Experimental): Systemically healthy subjects with periodontitis having interdental clinical attachment loss ≥ 3-5mm (stage II/III periodontitis) and probing pocket depth (PPD) ≥5mm (stage II/III periodontitis) and bleeding on probing ≥10% of sites.
  Interventions: Procedure: Non surgical periodontal therapy
- GROUP III: 40 coronary artery disease patients without periodontitis. (Experimental): Patients diagnosed with coronary artery disease with healthy periodontium having probing pocket depth (PPD)≤3mm, no clinical attachment loss (CAL=0) and bleeding on probing ≤ 10% of sites (CAD).
  Interventions: Procedure: Non surgical periodontal therapy
- GROUP IV: 40 periodontitis patients with coronary artery disease. (Experimental): Coronary artery disease (CAD) patients with periodontitis having interdental clinical attachment loss ≥3-5mm (stage II/III periodontitis) and probing pocket depth (PPD) ≥5mm (stage II/III periodontitis) and bleeding on probing ≥ 10%.
  Interventions: Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — Scaling and root planing is a deep cleaning below the gumline used to treat gum disease.
  Gum disease is caused by a sticky film of bacteria called plaque. Plaque is always forming on your teeth, but if they aren't cleaned well, the bacteria in plaque can cause your gums to become inflamed.
  Other Names: Scaling and root planing
  Arms: GROUP II: 40 periodontitis patients without coronary artery disease; GROUP III: 40 coronary artery disease patients without periodontitis.; GROUP IV: 40 periodontitis patients with coronary artery disease.

SUMMARY:
Untreated periodontal infection may result in transient bacteremia and toxaemia which may be the cause of adverse systemic events, leading to various systemic disorders. Amongst all the systemic diseases, cardiovascular disease has been recognized as a major systemic inflammatory condition that present similarities with periodontal disease. Increased systemic biomarkers of inflammation associated with periodontal disease have been interpreted as a mechanistic link between periodontitis and cardiovascular diseases.

Genetic factors are also known to play a pivotal role in influencing the inflammatory and immune response. Genetic polymorphisms are alterations in the DNA sequence found in general population. Most forms of periodontitis represent a life-long account of interactions between the genome and the environment. The previous literature has stated a strong association of genetic polymorphisms in periodontitis and coronary artery diseases. Identifying these polymorphisms can potentially lead to a better understanding of the mechanisms modulating the expression of inflammatory mediators as well as provides potential therapeutic targets in the prevention of periodontal disease. Two such novel polymorphisms have gained attention recently, namely the Dickkopf-3 and complement factor H polymorphisms.

Dickkopf-3 belongs to Dickkopf family of glycoproteins. Dickkopf-3 has been mainly investigated in oncology for its role as a tumor suppressor gene and as a therapeutic target in several types of human carcinomas. Recently, Dickkopf-3 gained attention as an emerging biomarker for cardiovascular and renal diseases. Dickkopf-3 has shown to play a role in pathophysiology of arterial wall thickening and abnormality implicated in atherosclerosis.

However, genetic polymorphism of Dickkopf-3 rs11544814 and complement factor H rs10737680 its protein levels have never been investigated in subgingival plaque samples of periodontitis patients with coronary artery disease specifically before and after non-surgical therapy. This may further improve our understanding of the influence of this polymorphism on the above mentioned systemic diseases.

DETAILED DESCRIPTION:
Periodontitis is a chronic immuno-inflammatory disease of the gingiva and supporting tissues which is initiated and perpetuated by key periodontal pathogens that results in the destruction of periodontal supporting structures and loss of alveolar bone, eventually culminating in tooth loss. It is further influenced by the complex interaction between periodontal pathogens and the host immune response. Untreated periodontal infection may result in transient bacteremia and toxaemia which may be the cause of adverse systemic events, leading to various systemic disorders. The presence of periodontal pathogens and their metabolic by-products in the oral cavity may get disseminated to the systemic circulation which may pose a risk for various systemic diseases such as cardiovascular disease, oral and colorectal cancer, gastrointestinal diseases, respiratory tract infection, adverse pregnancy outcomes, and diabetes.

Amongst all the systemic diseases, cardiovascular disease has been recognized as a major systemic inflammatory condition that present similarities with periodontal disease. Linking mechanisms between periodontal and cardiovascular disease include shared risk factors, increased fibrinogen, the role of white blood cells (WBC), the effect of bacterial lipopolysaccharide (LPS), and acute phase reactants such as C - reactive protein. Increased systemic biomarkers of inflammation associated with periodontal disease have been interpreted as a mechanistic link between periodontitis and cardiovascular diseases.

Although pathogenic bacteria and various other environmental factors are involved in pathogenesis of periodontitis, genetic factors are also known to play a pivotal role in influencing the inflammatory and immune response. Genetic polymorphisms are alterations in the DNA sequence found in general population. Most forms of periodontitis represent a life-long account of interactions between the genome and the environment. The previous literature has stated a strong association of genetic polymorphisms in periodontitis and coronary artery diseases. Identifying these polymorphisms can potentially lead to a better understanding of the mechanisms modulating the expression of inflammatory mediators as well as provides potential therapeutic targets in the prevention of periodontal disease. Two such novel polymorphisms have gained attention recently, namely the Dickkopf-3 and complement factor H polymorphisms.

Dickkopf-3 belongs to Dickkopf family of glycoproteins. This protein contains an N-terminal soggy domain and 2 conserved cysteine rich domains (CRDS) which is encoded by the Dickkopf-3 gene. These regulate the WNT signaling pathway, and other signaling cascades such as transforming growth factor beta (TGFβ) signaling. Dickkopf-3 has been mainly investigated in oncology for its role as a tumor suppressor gene and as a therapeutic target in several types of human carcinomas. Recently, Dickkopf-3 gained attention as an emerging biomarker for cardiovascular and renal diseases. Dickkopf-3 has shown to play a role in pathophysiology of arterial wall thickening and abnormality implicated in atherosclerosis. However, genetic polymorphism of Dickkopf-3 rs11544814 and its protein levels have never been investigated in patients with periodontitis with coronary artery disease. This may further improve our understanding of the influence of this polymorphism on the above mentioned systemic diseases.

Another novel polymorphism contributing to periodontitis and coronary artery disease is the complement factor H polymorphism. The complement pathway is an essential component of the innate immune system which participates in the elimination of pathogens and bridges the gap between innate and adaptive immunity. Complement factor H is a soluble complement regulator essential for controlling the alternative pathway in blood and on cell surfaces. By recognizing the host cell markers, complement factor H not only controls the complement during normal homeostasis, but also plays an important role by limiting complement mediated damage of diseased cells and tissues. Inadequate recognition of cells by complement factor H results in pathologies such as inherited atypical haemolytic uremic syndrome (aHUS), age related macular degeneration (ARMD), and membrano-proliferative glomerulonephritis type II. Recent studies reported that complement factor H polymorphism is associated with an increased risk of cardiovascular diseases in the elderly population. Studies have also been done to identify various complement factor H polymorphisms, however none of the studies have explored the role of complement factor H rs10737680 and its protein level in subjects with both periodontal disease and coronary artery disease occurring as a continuum. Its expression in periodontal tissues of cardiovascular disease patients is yet to be explored which might act as a potent health assessment tool associating periodontal and cardiovascular diseases in future.

NEED FOR THE STUDY While there are studies which have demonstrated the expression of Dickkopf-3 and complement factor H polymorphisms in various inflammatory conditions, there are no studies to state their expression in the subgingival plaque samples of periodontitis patients with coronary artery disease, specifically before and after non-surgical therapy. Also, the correlation of both these polymorphisms and their levels with periodontal and cardiac parameters has never been investigated so far. It is suggested that these polymorphisms may play a role as putative risk indicators in periodontitis subjects with coronary artery disease which may alter following non-surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Male and female patients within the age group of 30-65 years.
3. Patients having ≥ 10 remaining natural teeth.
4. No history of long term antibiotic use in past 6 months.

Exclusion Criteria:

1. Subjects with systemic conditions such as type I and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies/neoplasm and HIV infection will be excluded from the present investigation.
2. Subjects on drugs such as corticosteroids or antibiotics within 6 months of investigation or antiepileptic drugs (phenytoin or cyclosporine) having an impact on periodontal tissues will be excluded.
3. Pregnant women (pregnancy may alter the oral flora).
4. Current smokers and individuals who quit smoking less than 6 months.
5. Patients who have undergone periodontal therapy within the previous 6 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in periodontal parameters | Two years
  Change in Periodontal Probing Depth (measured in mm higher value indicate disease progression)
Change in periodontal variables | Two years
  Change in Clinical Attachment Level (measured in mm higher value indicate disease progression)
Change in periodontal criteria | Two years
  Change in Plaque Index (measured as a ratio, range: 0 to 3, maximum value indicates worse outcome and minimum value indicates better outcome )
Change in periodontal variables | Two years
  Change in Gingival index (measured as a ratio, higher value indicates severity of gingival inflammation
  )

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Meenakshi Ammal Dental college and hospital, Chennai, Tamil Nadu
  - Frontier lifeline Hospital, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng WL, Yang Y, Zhang XJ, Guo J, Gong J, Gong FH, She ZG, Huang Z, Xia H, Li H. Dickkopf-3 Ablation Attenuates the Development of Atherosclerosis in ApoE-Deficient Mice. J Am Heart Assoc. 2017 Feb 20;6(2):e004690. doi: 10.1161/JAHA.116.004690. PMID 28219919